CLINICAL TRIAL: NCT00002141
Title: A Phase I Trial to Evaluate the Safety and Pharmacokinetics of 1592U89
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Burroughs Wellcome (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 238A; 001
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1994-10

CONDITIONS: HIV Infections
Keywords: Biological Availability; Reverse Transcriptase Inhibitors; Food-Drug Interactions; abacavir
MeSH Terms: conditions — HIV Infections | interventions — abacavir

INTERVENTIONS:
Drug: Abacavir sulfate

SUMMARY:
To assess the safety of single oral doses of 1592U89 (abacavir succinate, ABC) administered to HIV-positive individuals. To determine the pharmacokinetics of 1592U89 after single oral doses. To determine the effects of food on the bioavailability of 1592U89.

DETAILED DESCRIPTION:
Patients are randomized in a double-blinded manner, with 12 patients entering the treatment arm and 6 patients entering the control arm. Patients in the treatment arm receive 6 single escalating doses of 1592U89 separated by at least a 6-day washout period. Patients in the control arm receive 6 single oral doses of placebo at least 6 days apart. The second and third doses of 1592U89 are equivalent. During these doses, investigators study the effects of food on the pharmacokinetics of 1592U89 by giving half of the patients the second dose with a standardized, high-fat breakfast and giving the other half the dose in a fasted state. During the third dose, patients are crossed over so that patients who received the second dose with a meal now receive it in a fasted state, and vice versa. Following the sixth dose, investigators break the blind. Patients who received 1592U89 take a seventh dose in solution form and return for follow-up at least 7 days later; patients who received placebo receive no further treatment or follow-up. Serial blood and urine samples are collected before and after each administration of 1592U89 (or placebo) for determination of plasma and urine concentrations of 1592U89, and investigators monitor patients closely for adverse events or abnormal laboratory test findings.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* HIV infection, as documented by ELISA/Western blot detection of HIV antibody, positive p24 antigen assay, positive viral culture, or other accepted technique.
* Written informed consent of parent or legal guardian if under age 18.

Exclusion Criteria

Co-existing Condition:

Excluded:

* Debilitating disease, as a result of HIV or associated therapies, that, in the opinion of the investigator, might prevent the patient from completing 6-week dosing period.
* Malabsorption syndrome or other gastrointestinal dysfunction that might interfere with drug absorption.

Concurrent Medication:

Excluded:

* Prescription or over-the-counter medication that cannot be withheld for 48 hours prior to dosing and during the 6 dosing periods. (Note:
* Antiretrovirals must be withheld for 24 hours prior to dosing and during the day of dosing.)
* Other investigational treatments (treatments available through a Treatment IND or other expanded access mechanism is evaluated individually in consultation with the sponsor).
* Alcoholic beverages within 48 hours before dosing and during the day of dosing.
* Coffee, tea, and other xanthine-containing beverages and foods on the day of dosing.

Patients with the following symptoms or conditions are excluded:

History of hepatitis, pancreatitis, or cardiomyopathy within the last 5 years.

Risk Behavior:

Excluded:

Current alcohol or illicit drug use that might interfere with the patient's ability to comply with the dosing schedule and protocol evaluations, as determined by the investigator.

Ages: 13 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18
Dates: Start 1994-07

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Georgetown Univ Med Ctr, Washington D.C., District of Columbia
  - Ctr for Phase I Research, Wichita, Kansas